CLINICAL TRIAL: NCT03153072
Title: Evaluation of the Pharmacokinetic Profile, Pharmacodynamic Effects, Acceptability and Tolerability of an Oral Amiodarone Solution of 15 mg / mL in Children With Supra Ventricular Tachycardia
Acronym: Enteramio
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: decision of the investigator
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0020
Record Dates: First submitted 2017-04-28; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A child with supraventricular tachycardia (Other)
  Interventions: Biological: Assess the absorption of oral amiodarone

INTERVENTIONS:
Biological: Assess the absorption of oral amiodarone — Evaluate the pharmacokinetics of oral amiodarone solution at 15 mg / mL after oral administration

SUMMARY:
The supra ventricular tachycardia is the most common symptomatic arrhythmia in pediatrics. Amiodarone is an antiarrhythmic drug used in this indication. Pharmacokinetic, efficacy and safety data are not known in the pediatric population due to the lack of a suitable specialty available on the market.

The development of an amiodarone oral solution formulation adapted to this age group should provide a therapeutic alternative and collect data on the pharmacokinetics, efficacy, acceptability and tolerability of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Child (boy or girl) with supra ventricular tachycardia diagnosed by ECG recording.
* Child aged 0 to 11 years.
* Child whose parents / legal representative (s) agree to sign a consent form.
* Child whose opinion / agreement has been / has been attempted to be collected.
* Child and parents / legal representative (s) being ready and able to participate in the study, understanding and committing to respect the procedures of the study throughout its duration.
* Child enrolled in a social security scheme.
* Child with a body mass index between the 3rd and the 97th percentile.

Exclusion Criteria:

* A child with a known hypersensitivity to the active ingredient, iodine or any of the excipients of the study formulation.
* Child who has already been treated with amiodarone (as a capsule or with the oral injectable form)
* Impossibility of taking blood samples.
* Hyperthyroidism (TSH <laboratory low standard).
* Disruption of liver function (ASAT> 3N and / or ALT> 3N).
* Renal impairment (Cl creat <30 mL / min)
* Hepatic insufficiency (TP or factor V <70%)
* Inotropic support.
* Uncorrected severe ionic disorders.
* Extension of the QTc space before the implementation of the treatment (> 450 ms).
* Non-paired sinus disease.
* Concomitant treatment with a drug which has an absolute contraindication with amiodarone.
* Child with gastrointestinal disorders such as malabsorption syndrome.
* Weight <2.5 kg.
* Child whose mother was treated with amiodarone during pregnancy.
* Child who received another product under investigation or participated in another study within 60 days of the start of this study.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Blood analysis of the absorption of oral amiodarone solution in a child with supraventricular tachycardia | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France